CLINICAL TRIAL: NCT00108810
Title: Randomized, Double-Blind, Parallel, Placebo Controlled 4 Week Proof-of-Concept Study to Evaluate the Safety and Efficacy of Transdermal Ketoprofen When Administered With Controlled Heat in Patients With Mild to Moderate OA Pain of the Knee
Brief Title: Transdermal Ketoprofen to Treat Mild to Moderate Osteoarthritis (OA) Pain of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZMK-202
Record Dates: First submitted 2005-04-18; First posted 2005-04-19 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-05

CONDITIONS: Pain; Osteoarthritis, Knee
Keywords: Pain; Osteoarthritis; OA; Mild to Moderate Osteoarthritis (OA) Pain of the Knee
MeSH Terms: conditions — Pain; Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transdermal Ketoprofen Patch with CHADD (Experimental)
  Interventions: Drug: Transdermal Ketoprofen Patch with CHADD
- Placebo patch and a dummy heating unit (Placebo Comparator)
  Interventions: Drug: Placebo transdermal patch

INTERVENTIONS:
Drug: Transdermal Ketoprofen Patch with CHADD — 12 hours patch application for 28 days
  Other Names: Matrix Transdermal Ketoprofen/CHADD Sytem
  Arms: Transdermal Ketoprofen Patch with CHADD
Drug: Placebo transdermal patch — 12 hours application for 28 days
  Other Names: Placebo patch with dummy heating unit
  Arms: Placebo patch and a dummy heating unit

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the investigational ketoprofen patch with a controlled heating patch, compared to placebo (inactive substance) for the treatment of pain caused by osteoarthritis.

DETAILED DESCRIPTION:
Proof-of-concept study, multicenter, randomized, double-blind, parallel-group, placebo-controlled study designed to evaluate the safety and efficacy of a transdermal ketoprofen patch with CHADD heat versus a placebo patch with dummy heat in patients with mild to moderate pain associated with osteoarthritis of the knee. After screening, patients discontinue all analgesic medication (except ≤325 mg aspirin daily for cardioprotective purposes). Patients selected a target knee (right or left), and all efficacy evaluations were completed with respect to this target knee. After discontinuing analgesics for at least 48 hours, and when the average pain intensity over the previous 24 hours for the target knee was ≥40 mm using a 100 mm visual analog scale (VAS), patients were randomized in a 1:1 fashion to receive treatment with either the transdermal ketoprofen patch with CHADD heat or the placebo patch with dummy heat. Patients treated the target knee each night for 12 hours (± 1 hour) for 4 weeks. Patients returned to the study site every 7 days (± 1 day) for study evaluations. Throughout the study, patients were allowed to take up to 2000 mg acetaminophen per day as rescue medication; however, rescue medication was not allowed within the 48 hours prior to efficacy evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between forty (40) and seventy-five (75) years of age.
* Patient has clinically diagnosed radiographic evidence of osteoarthritis of the knee within the past year.

Exclusion Criteria:

* Patient has known allergy to nonsteroidal anti-inflammatory drugs (NSAIDs) (including aspirin) or has a suspected hypersensitivity, allergy or other contraindication to any compound present in the study medication.
* Patient has a history of significant gastrointestinal disease or previous gastrointestinal upset following NSAID administration.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2005-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the WOMAC pain subscale score | 28 days

SECONDARY OUTCOMES:
Number of participants wih adverse events | 28 days
Patient Global Satisfaction score | 28 days
  Patient global satisfaction score at Study Visit 5
Mean change from baseline for average pain over the last 24 hours VAS scores | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: David Borenstein, MD, Principal Investigator — The Center for Rheumatology; H F Farmer, MD, Principal Investigator — Radiant Research Inc.; Larry Gilderman, DO, Principal Investigator — University Clinical Research; Soledad Lee, MD, Principal Investigator — Southbay Pharma Research; Joseph A Markenson, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (5):
- United States (5):
  - SouthBay Pharma Research, Buena Park, California
  - The Center for Rheumatology and Bone Research, Washington D.C., District of Columbia
  - Radiant Research, Daytona Beach, Florida
  - University Clinical Research, Pembroke Pines, Florida
  - Hospital for Special Surgery, New York, New York